CLINICAL TRIAL: NCT00002292
Title: Inhaled Versus Intravenous Pentamidine in Pneumocystis Carinii Pneumonia in the Acquired Immunodeficiency Syndrome
Brief Title: A Study of Two Forms of Pentamidine in the Treatment of Pneumocystis Carinii Pneumonia (PCP) in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LyphoMed (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 023B; 88-001
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-08

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Pentamidine; Injections, Intravenous; Administration, Inhalation; Aerosols; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Respiratory Aspiration; Acquired Immunodeficiency Syndrome | interventions — Pentamidine

INTERVENTIONS:
Drug: Pentamidine isethionate

SUMMARY:
To compare parenteral versus inhaled pentamidine in patients with documented Pneumocystis carinii pneumonia (PCP) with AIDS.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Previous history of adverse reaction to pentamidine.
* History of asthma.
* Pulmonary Kaposi's sarcoma.

Patients with the following are excluded:

* Previous history of adverse reaction to pentamidine.
* History of asthma.
* Pulmonary Kaposi's sarcoma.
* Inability to understand the consent procedure.

All patients hospitalized at Cedars-Sinai Medical Center with AIDS and possible Pneumocystis carinii pneumonia (PCP) will be eligible.

* Patients with HIV antibody or AIDS and a clinical presentation suggesting PCP are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- LyphoMed Inc, Rosemont, Illinois, United States

REFERENCES:
- [Background] Soo Hoo GW, Mohsenifar Z, Meyer RD. Inhaled or intravenous pentamidine therapy for Pneumocystis carinii pneumonia in AIDS. A randomized trial. Ann Intern Med. 1990 Aug 1;113(3):195-202. doi: 10.7326/0003-4819-113-3-195. PMID 2197910
- [Background] Conte JE Jr, Chernoff D, Feigal DW Jr, Joseph P, McDonald C, Golden JA. Intravenous or inhaled pentamidine for treating Pneumocystis carinii pneumonia in AIDS. A randomized trial. Ann Intern Med. 1990 Aug 1;113(3):203-9. doi: 10.7326/0003-4819-113-3-203. PMID 2197911